CLINICAL TRIAL: NCT05647603
Title: Role of Parents Concerning Information of Adolescents About Contraception
Acronym: Info-Contra
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_014_Info-Contra
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Parents of Adolescent
Keywords: adolescents; contraception; information
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group "Parents of adolescents": Parents of adolescents aged 12 to 18
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Information about contraception

SUMMARY:
Adolescence is a period of intensive physical and psychological changes, with notably the start of sexuality. During this period of sexual discovery, a lack or a misuse of contraception may be responsible for unwanted pregnancy.

So, sexual education and information about contraception are crucial. Teenagers often consult Internet or discuss with friends to have information but they can be not true or precise. They can also consult health professionals, however shyness and fear can hold them back. Information about contraception may also be given by their parents. The physical closeness and the trust that adolescents have in their parents can promote dialogue.

DETAILED DESCRIPTION:
the aim of the study is to describe information about contraception given by parents to adolescents

ELIGIBILITY:
Inclusion Criteria:

* Parents (father or mother) of adolescents (boy or girl) aged 12 to 18
* agreeing to participate to the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of adolescents aged 12 to 18
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Definition of contraception | Day 0
  Parents have explained or not that contraception is all methods aimed at reversibly preventing an unwanted pregnancy
Contraception methods | Day 0
  Parents have explained or not all contraception methods (condom for man, condom for woman, control pills, contraceptive implant, intra-uterine device, contraceptive patch, contraceptive ring, spermicide

CONTACTS AND LOCATIONS:
Overall Officials: Lapree Lucie, Principal Investigator — Université de Reims Champagne-Ardenne
Locations (1):
- Université de Reims Champagne Ardenne, Reims, France